CLINICAL TRIAL: NCT00477880
Title: Treatment of Ménétrier's Disease With EGF Receptor Blockade
Brief Title: Cetuximab in Treating Patients With Ménétrier Disease at High Risk of Developing Stomach Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert J. Coffey, Asst Professor, Otolaryngology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000546501; P30CA068485 (NIH); VU-VICC-GI-0602; VU-VICC-IRB-000851; NCT00268736 (obsolete NCT alias)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Cancer; Precancerous Condition
Keywords: gastric cancer; giant hypertrophic gastritis
MeSH Terms: conditions — Stomach Neoplasms; Precancerous Conditions; Gastritis, Hypertrophic | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab (Experimental): Cetuximab lV weekly at an initial loading dose of 400 ml/m2, followed by three weekly maintenance doses of 250 mg/m2. Four infusions of C225 will be defined as a course of therapy.
  Interventions: Biological: Cetuximab

INTERVENTIONS:
Biological: Cetuximab
  Other Names: C225

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This clinical trial is studying how well cetuximab works in treating patients with Ménétrier disease at high risk of developing stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate clinical and biochemical parameter response in patients with Ménétrier disease at high risk of developing gastric cancer treated with cetuximab.

OUTLINE: This is a non-randomized study.

Patients receive cetuximab IV on days 1, 8, 15, and 22. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients complete a quality of life questionnaire at baseline and during week 4.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Ménétrier disease

  * Symptomatic disease, including gastrointestinal symptoms which interfere with daily life

    * Patient is considering surgery
* Must have failed medical therapy that was given for 6 months
* No Helicobacter pylori infection

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No NYHA class III-IV cardiovascular disease
* No clinically unstable pulmonary disease
* No chronic disease requiring ongoing therapy for stabilization, including any of the following:

  * Uncontrolled diabetes mellitus
  * Malignancy
  * Thyroid disease
  * Hypertension
  * Active infections requiring systemic antibiotics, antivirals, or antifungals
  * Uncontrolled seizure disorder
  * Active neurological disease
* No unstable coagulation disorders (e.g., hemorrhagic diatheses or active bleeding disorders) that require medical management

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2001-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Response | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Coffey, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee